CLINICAL TRIAL: NCT02821858
Title: A Phase 1, Double-blind, Placebo-controlled, Randomized, Single Ascending Dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of Odalasvir and AL-335 in Healthy Japanese Subjects
Brief Title: Study to Investigate the Pharmacokinetics, Safety and Tolerability of Odalasvir and AL-335 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108178; 64294178HPC1005 (Other: Janssen Research & Development, LLC); 2015-005639-42 (EudraCT Number)
Record Dates: First submitted 2016-06-10; First posted 2016-07-04 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Healthy
MeSH Terms: interventions — odalasvir; adafosbuvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (6):
- Panel 1: Treatment A (Experimental): Participants will receive odalasvir (ODV) 50 milligram (mg) (n=8) or placebo (n=2) on Day 1.
  Interventions: Drug: Odalasvir (ODV); Drug: Placebo
- Panel 1: Treatment B (Experimental): Participants will receive ODV 100 mg (n=8) or placebo (n=2) on Day 1.
  Interventions: Drug: Odalasvir (ODV); Drug: Placebo
- Panel 1: Treatment C (Experimental): Participants will receive ODV 300 mg (n=8) or placebo (n=2) on Day 1.
  Interventions: Drug: Odalasvir (ODV); Drug: Placebo
- Panel 2: Treatment D (Experimental): Participants will receive AL-335 400 mg (n=8) or placebo (n=2) on Day 1 of Period 1. Each treatment period will be separated by a washout period of 7 days.
  Interventions: Drug: AL-335; Drug: Placebo
- Panel 2: Treatment E (Experimental): Participants will receive AL-335 800 mg (n=8) or placebo (n=2) on Day 1 of Period 2. Each treatment period will be separated by a washout period of 7 days.
  Interventions: Drug: AL-335; Drug: Placebo
- Panel 2: Treatment F (Experimental): Participants will receive AL-335 1,200 mg (n=8) or placebo (n=2) on Day 1 of Period 3. Each treatment period will be separated by a washout period of 7 days.
  Interventions: Drug: AL-335; Drug: Placebo

INTERVENTIONS:
Drug: Odalasvir (ODV) — ODV 50 mg (1 tablet) in Treatment A, 100 mg (2 tablets of 50 mg) in Treatment B and 300 mg (6 tablets of 50 mg) in Treatment C.
  Arms: Panel 1: Treatment A; Panel 1: Treatment B; Panel 1: Treatment C
Drug: AL-335 — AL-335 400 mg (1 tablet) in Treatment D, 800 mg (2 tablets of 400 mg) in Treatment E and 1200 mg (3 tablets of 400 mg) in Treatment F.
  Arms: Panel 2: Treatment D; Panel 2: Treatment E; Panel 2: Treatment F
Drug: Placebo — Matching placebo will be administered.

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics (PK), safety and tolerability following single oral administration of ascending doses of odalasvir (ODV) in healthy Japanese participants (Panel 1) and to investigate the PK, safety and tolerability following single oral administration of ascending doses of AL-335 in healthy Japanese participants (Panel 2; Sequential Design).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a Japanese participant who has resided outside Japan for no more than 5 years and whose parents and grandparents are Japanese as determined by participant's verbal report
* Participant must have a body mass index (BMI: weight in kilogram [kg] divided by the square of height in meters) of 18.0 to 30.0 kilogram per meter square (kg/m^2), extremes included and a body weight not less than 50.0 kilogram (kg)
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening. If there are abnormalities, the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the Investigator
* Participant must have a blood pressure (after the participant supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted
* Female participant must agree to not donate eggs (ova, oocytes) for the purpose of assisted reproduction during the study and for a period of 60 days (Panel 1) or 30 days (Panel 2) after study drug administration or until the last follow-up visit, whichever occurs later

Exclusion Criteria:

* Participant has a history of liver or renal insufficiency (estimated creatinine clearance below 80 milliliters per minute [mL/min]); significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the Investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic or metabolic disturbances
* Participant has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant with a past history of heart arrhythmias (for example, extra systolic beats or tachycardia at rest); risk factors associated with Torsade de Pointes such as hypokalemia or family history of short/long QT syndrome or sudden unexplained death (including sudden infant death syndrome) in a first-degree relative [for example, sibling, offspring, or biological parent])
* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participant has known allergies, hypersensitivity, or intolerance to odalasvir (ODV) or AL-335 or its excipients

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Odalasvir (ODV) | From Day 1 to Day 14 after intake of ODV
  The Cmax is the maximum observed analyte concentration.
Time to Reach Maximum Observed Concentration (Tmax) of ODV | From Day 1 to Day 14 after intake of ODV
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUClast) of ODV | From Day 1 to Day 50-55 after intake of ODV
  The (AUC [0-last]) is the area under the analyte concentration-time curve from time 0 to time of the last quantifiable concentration.
Elimination Rate Constant (Lambda[z]) of ODV | From Day 1 to Day 50-55 after intake of ODV
  Lambda(z) is first order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Elimination Half-Life (t1/2) of ODV | From Day 1 to Day 50-55 after intake of ODV
  Elimination half-life (t[1/2]) is associated with the terminal slope (lambda [z]) of the semi-logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Area Under the Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of ODV | From Day 1 to Day 50-55 after intake of ODV
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability for ODV | Up to 50-55 days after intake of ODV
Maximum Observed Concentration (Cmax) of AL-335 | From Day 1 to Day 4 after intake of AL-335
  The Cmax is the maximum observed analyte concentration.
Time to Reach Maximum Observed Concentration (Tmax) of AL-335 | From Day 1 to Day 4 after intake of AL-335
  The Tmax is defined as actual sampling time to reach maximum observed concentration.
Area Under the Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUClast) of AL-335 | From Day 1 to Day 4 after intake of AL-335
  The (AUC [0-last]) is the area under the concentration-time curve from time 0 to time of the last quantifiable concentration.
Elimination Rate Constant (Lambda[z]) of AL-335 | From Day 1 to Day 4 after intake of AL-335
  Lambda(z) is first order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Elimination Half-Life (t1/2) of AL-335 | From Day 1 to Day 4 after intake of AL-335
  Elimination half-life (t[1/2]) is associated with the terminal slope (lambda [z]) of the semi-logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Area Under the Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of AL-335 | From Day 1 to Day 4 after intake of AL-335
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability for AL-335 | Up to 30 to 35 days after last intake of AL-335

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Developement, LLC Clinical Trial, Study Director — Janssen Research and Developement, LLC
Locations (1):
- Surrey, United Kingdom